CLINICAL TRIAL: NCT01448122
Title: A Randomized, Single-blind Study of the Ability of Avène Compact Honey to Prevent Pigmentation Induced by Visible Light in Subjects With Skin Phototype III or IV
Brief Title: Avene Compact Honey for Prevention of Pigmentation From Visible Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Principal Investigator, Dr Robert Bissonnette, Robert Bissonnette MD, FRCPC, Pierre Fabre Dermo Cosmetique
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RV 4140 A 2011 176
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Prevention of pigmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Avene Compact Honey SPF 50 (Active Comparator): Study product will be scraped from compact case and weighed. Product will be applied to half the area to be exposed with visible light at a concentration of 2 mg/mL.
  Interventions: Other: Avene Compact Honey SPF 50
- No intervention (No Intervention): Half of the area to be exposed to visible light will have no study product applied.

INTERVENTIONS:
Other: Avene Compact Honey SPF 50 — Patients will have part of their back covered with 2 mg/mL of Avene Compact Honey SPF 50.
  Other Names: Avene Compact Doré SPF 50
  Arms: Avene Compact Honey SPF 50

SUMMARY:
The main objective of the study is to assess the efficacy of Avène Compact Honey in preventing pigmentation induced by visible light in subjects with a phototype III or IV.

Patients will be exposed to a range of visible light to areas on the back to confirm study eligibility. Patients showing pigmentation after 7 days on the exposed areas will be eligible to continue.

Eligible patients will have study product applied to part of the back. The back will be exposed to a range of light based on the minimum exposure inducing pigmentation previously ascertained. The area where study product is applied will have a higher range of light exposure than the area without the study product.

Seven days later, the areas will be examined to determine the lowest exposure inducing pigmentation on the sides with and without study product. The color will also be measured between two identical exposures with and without the applied study product.

DETAILED DESCRIPTION:
Part A At Day -7, all subjects will be exposed to a range of doses of visible light on an approximately 0.90 cm diameter area on the back to ascertain their predisposition for pigmentation induced by visible light. The doses will be 30, 40, 60, 80, 100 and 120 J cm-2. At the Day 0 visit, subjects' pigmentation will be determined by investigator visual assessment. Subjects with a lowest observed pigmentation at the 30 J cm-2 or the 120 J cm-2 dose will not continue in the study. For each subject that continues, the area where Avène Compact Honey will be applied on the back will be randomized. At least 15 minutes later, unprotected areas will be exposed to doses ranging from ~1/20th to 1.8 times the lowest dose of visible light that induced pigmentation at Day -7. To not unnecessarily over expose subjects, the first 3 will have protected areas exposed to doses ranging from ~half to 16 times the lowest dose of visible light that induced pigmentation at Day -7. All subjects will have an additional exposure on the protected side equal to the highest dose of the unprotected side for colorimetric comparison. Subjects will be examined at Day 7 (seven days after visible light exposure). Pigmentation on all exposed areas will be evaluated by investigator visual assessment. The colorimetric measurements on protected and unprotected skin will be recorded for the equivalent exposures and for adjacent skin. The exposed area on the protected side to be tested with colorimetric analysis will be hidden during the investigator visual assessment. The minimum dose on the unprotected side and an area of unprotected and unexposed skin will be hidden from the colorimetric evaluator to maintain the blind. The lowest visible light dose inducing pigmentation will be recorded for both the unprotected and protected areas. If the first three subjects are only pigmented at either the 16X level or not at all on the protected side, then the remaining subjects in the study will be exposed at doses ranging from 0.7 to as high as 24 times the lowest dose of visible light that induced pigmentation at Day -7.

Part B At Day 0, all subjects will be exposed to a range of doses of visible light on an approximately 0.90 cm diameter area on the back to ascertain their disposition for pigmentation induced by visible light. The doses will be 8, 40, 80, 160, 320 and 480 J cm-2. At the Day 7 visit, subjects' pigmentation will be determined by investigator visual assessment. Subjects will be divided into 2 cohorts. Cohort A will contain 5 subjects of phototype IV with dark skin and cohort B will contain 5 subjects with skin phototype V.

Part C At Day -7, all subjects will be exposed to a range of doses of visible light on an approximately 0.90 cm diameter area on the back to ascertain their predisposition for pigmentation induced by visible light. The doses will be 8, 40, 80, 160, 320 and 480 J cm-2. At the Day 0 visit, subjects' pigmentation will be determined by investigator visual assessment. Subjects with a lowest observed pigmentation at the 8 J cm-2 dose will not continue in the study and neither will subjects showing no pigmentation at 480 J cm-2. For each subject that continues, the area where Avène Compact Honey will be applied on the back will be randomized and then receive the application. At least 15 minutes later, protected areas will be exposed to doses of 32, 160, 320, 640, 1280 and 1920 cm-2. Unprotected areas will be exposed to the same doses as Day 0. To not unnecessarily over expose subjects, those with a lowest observed pigmentation at Day 0 of 40 or 80 J cm-2 will have the maximum exposure at Day 0 determined at the investigators discretion. Subjects will be examined at Day 7 (seven days after visible light exposure). Pigmentation on all exposed areas will be evaluated by investigator visual assessment. The lowest visible light dose inducing pigmentation will be recorded for both the unprotected and protected areas. The colorimetric measurements on protected and unprotected skin will be recorded for the equivalent exposures and for adjacent skin. Four areas of unprotected and protected skin will be hidden from the colorimetric evaluator to maintain the blind. Subjects will be divided into 2 cohorts. Cohort A will contain 5 subjects of phototype IV with dark skin and cohort B will contain 5 subjects with skin phototype V.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 18 years of age or older at time of consent.
2. Subject has a skin phototype of III or IV.
3. Subject (or subject's partner), male or female, is willing to use effective contraceptive method for at least 30 days before Day -7 and until Day 7. Effective contraceptive methods are:

   1. Barrier methods such as condom, sponge or diaphragm combined with spermicide in foam, gel or cream;
   2. Hormonal contraception (oral, intramuscular, implant or transdermal) which include Depo-Provera, Evra and Nuvaring;
   3. Intrauterine device (IUD);
   4. Sterilization such as tubal ligation, hysterectomy or vasectomy;
   5. Postmenopausal state for at least 1 year for female subject or female partner of male subject;
   6. Same-sex partner;
   7. Abstinence.
4. Subject must be willing to avoid exposure to UV radiation (tanning beds, phototherapy, and sunlight) on the back for the duration of the study.
5. Subject is capable of giving informed consent and the consent must be obtained prior to any study related procedures.
6. Subject has sufficient pigmentation at Day 0 in at least one area after exposure to varying doses of visible light at Day -7.

Exclusion Criteria:

1. Subject is currently pregnant or lactating.
2. Subject has a known allergy to the study product or a component of the study product.
3. Subject has used photosensitizing medication (in UV and in the visible range) within 30 days of the Day -7 visit up to the Day 7 visit.
4. Subject has a history of photodermatosis.
5. Subject has the presence of a skin disorder in the area to be irradiated that would either put the subject at increased risk or interfere with pigmentation evaluation.
6. Subject has a medical condition or is taking medication that could put him or her at undue risk.
7. Subject has a cardiovascular, pulmonary, digestive, neurological, urinary, psychiatric, hematological, immunological, or endocrinal pathology that is unstable or able to interfere with the study.
8. Subject has undergone organ removal or organ transplant
9. Subject is currently receiving treatment that may interfere with interpretation of the study results.
10. Subject for whom, in the Investigator's opinion, pigmentation on the back will be difficult to evaluate (such as subjects with excessive hair or a tattoo).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Lowest mean fluence inducing visible pigmentation | 7 days
  Lowest mean fluence inducing visible pigmentation 7 days after visible light exposure for skin protected with Avène Compact Honey as compared to unprotected skin.

SECONDARY OUTCOMES:
Mean difference in pigmentation darkness | 7 Days
  Mean difference in pigmentation (as evaluated by the L* component of colorimetric measurements) between exposed and non exposed skin according to fluence for skin protected with Avène Compact Honey as compared to unprotected skin.
Adverse Events | 7 Days
  The safety of Avène Compact Honey measured by the number of adverse events and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, FRCPC, Principal Investigator — Innovaderm Research Inc.
Locations (1):
- Innovaderm Research Inc, Montreal, Quebec, Canada